CLINICAL TRIAL: NCT02066441
Title: The Effect of Vitamin D on Serum Vitamin D Levels, Bone Formation, Resorption, and Mineral Density, Inflammation, Flexibility, and Balance in the Elderly
Brief Title: Vitamin D's Effect on Physical Performance in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Biotics, Inc. (Industry)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20120195
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Family Member
Keywords: Vitamin D; bone formation; resorption; mineral density; inflammation; flexibility; balance; elderly
MeSH Terms: conditions — Inflammation | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-D-Mulsion Forte® (Experimental): Bio-D-Mulsion Forte® at a dosage level of 2 drops (4,000 IU) once daily for the 6-month treatment period.
  Interventions: Dietary Supplement: Bio-D-Mulsion Forte®
- Placebo (Placebo Comparator): Placebo a dosage level of 2 drops once daily for the 6-month treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bio-D-Mulsion Forte® — According to the company's literature, Bio-D-Mulsion Forte® contains: vitamin D (as cholecalciferol), a water and gum Arabic emulsifier base, and sesame oil. This product is documented online at the following web address: http://www.bioticsresearch.com/node/1570
  Arms: Bio-D-Mulsion Forte®
Other: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare vitamin D deficient and vitamin D sufficient elderly individuals and examine the effect of a vitamin D dietary supplement on serum vitamin D level, bone formation, resorption, and mineral density, flexibility, balance, general inflammation,and quality of life. Enhancing nutritional status is necessary to prevent the continued proliferation of chronic diseases, e.g., bone disease and other chronic disorders thought to now be related to low levels of vitamin D, which are some of the leading disablers and killers of Americans. Americans also have difficulties with compliance to prescription medications due to their toxicity and side effects. This study aims to learn more about how a vitamin D nutritional supplement may improve nutritional status and enable the body to normalize system functioning,which may improve the quality of life for people with vitamin D deficiency. The results of this research will be used to determine if vitamin D is beneficial for overall health among elderly individuals.

DETAILED DESCRIPTION:
The proposed study has two parts and is observational (first part) and experimental (second part) in design. The purpose of the first part of this study is a cross-sectional investigation of the relationship among vitamin D status, vitamin D intake and sun exposure, and physical performance in 130 community dwelling older adult (≥55 years old). The purpose of the second part of the study is a 6-month, randomized, double-blind, placebo-controlled trial to evaluate the effect of vitamin D supplementation (Bio-D-Mulsion Forte®) for improving physical performance, serum levels of 25-OH-vitamin D, PTH, bone formation (osteocalcin), bone resorption (type 1 cross linked C telopeptide (CTX)), and bone mineral density (dual energy x-ray absorptiometry in a sub-sample of 20 participants) in 40 participants (≥55 years of age) who are vitamin D insufficiency at baseline (<30 ng/ml serum 25(OH)D). Secondary outcomes will include body composition, lower back/hamstring flexibility, balance, gustatory response to the treatment, general inflammation, quality of life, depression, fear of falling, history of falls, and food security. Information on sun exposure, vitamin D and calcium intake, physical activity level, and reflectance calorimetry will also be collected. Participants will be assessed at baseline and 6-months follow-up. This part of the study will consist of two treatment arms: (a) vitamin D dietary nutritional supplement and (b) placebo.

The primary risk for the placebo group is that they will show no improvement in serum levels of 25-OH-vitamin D, bone formation, bone resorption, bone mineral density, and secondary outcomes associated with vitamin D supplementation. However, they are not being restricted in any way to receive vitamin D through sunlight exposure and their food. Each participant in the placebo group will also receive a 6-month supply of the vitamin D supplement (Bio-D-Mulsion Forte®) at the conclusion of their participation in the study. Additionally, the risk of placebo is also offset by the knowledge gained from actually receiving a serum level 25-OH-vitamin D score at baseline and 6-months follow-up, which is not typically assessed by the average provider. Finally, the short-term period of the study does not increase long-term health risks associated with the study, as other studies have utilized placebo-controlled trials with vitamin D deficient adults previously and have observed no adverse effects . Normal serum levels of 25-OH-vitamin D can be achieved within 2-5 months according to the literature.

The health risks associated with consuming a vitamin D dietary supplement are inconclusive. Hypercalcemia is one potential adverse effect, but according to one review no increases in mean calcium levels occurred with higher vitamin D intakes tested in controlled trials up to 100,000 IU per day. For single cases of hypercalcemia from randomized controlled trials, cases of mild hypercalcemia were reported in 2 of 28 studies, which resolved on repeating fasting samples in one study and were actually more frequent in the placebo group in the other study. Additionally, hypercalcemia has been mostly found in cases of persons with serum levels of 25(OH)D greater than 240 nmol/L.

An increased risk of nephrolithiasis was found in one randomized controlled trial (the Women's Health Initiative (WHI)), which tested 400 IU vitamin D in combination with 1000 mg of calcium. The reason for nephrolithiasis in this study is unclear; factors include: (1) this study may have been large enough to detect a small risk of nephrolithiasis with vitamin D supplementation; (2) nephrolithiasis was caused by the calcium supplement intake taken in combination with the vitamin D as part of the protocol; and/or (3) the nephrolithiasis was caused by the additional calcium and vitamin D supplements taken by the majority of participants outside the study protocol. The low dose of vitamin D used in the WHI argues against a causal role of the increased risk of nephrolithiasis. Based on epidemiologic data, a higher vitamin D intake was not independently associated with nephrolithiasis in one large cohort consistent with findings from a recent study of 18 healthy postmenopausal women with vitamin D deficiency where vitamin D supplementation did not increase urinary calcium excretion. On the other hand, calcium supplementation was associated with a 20% increased risk of nephrolithiasis in the Nurses Health Study I.

The issue of vascular calcification has also been noted as a potential risk of vitamin D supplementation. However, reports in the literature continue to be restricted to extremely high doses of vitamin D3 or administration of the active hormonal form, 1,25(OH)2D3 and/or related analogues, and most of these reports are in animals, not humans. No credible evidence exists to support the notion that oral vitamin D doses up to and even exceeding 10,000 IU per day are associated with vascular calcification in humans, including dialysis patients, and no basis exists for identifying vascular calcification as a critical effect.

Participants may experience discomfort while answering the questionnaires and while undergoing the venipuncture, but they may stop the assessments at any time. Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the IRB.

The vitamin D dietary supplement should be harmless without any food allergy or sensitivity. No episodes of side effects have been reported to Biotics Research Corporation, the manufacturer, by consumers in the previous 5 years.

A toxicology search for each component reveals no unique toxicity characteristic of the materials. As reported by Biotics Research Corporation, thousands of people currently use Bio-D-Mulsion Forte®, and Biotics Research Corporation is unaware of significant toxicities. A major concern with raw natural products is the presence of contaminants.

Biotics Research Corporation operates in accordance with D-SHEA regulations, and Bio-D-Mulsion Forte® is made of the highest purity, quality, and potency. Biotics Research Corporation manufacturers their products under strict GMP guidelines in an FDA-registered facility, is licensed by the Texas Department of State Health Services Regulatory Licensing Unit as a Food and Non-prescription Drug Manufacturer, and is licensed by Health Canada (Site License) and is considered to be in compliance with the GMP requirements of their Natural Health Products Regulations. Biotics Research Corporation conducts multiple quality control tests on all of its products.

Participants will incur no additional appreciable psychological or social risks by participating in this study, although they may undergo psychological and physical discomfort sometimes. The process of interviewing during the assessment may cause discomfort. Discomfort or fatigue may also be experienced in completing the assessment battery.

Alternatives to this study include prescription medications, sun exposure, exercise, dietary modification, and other nutritional supplements. The risks of medications can be very significant, including life-threatening, but the risk of taking nutritional supplements is not totally understood, since they are not regulated by the FDA. Medications and nutritional supplements, as part of a change in lifestyle behaviors, may also prove to be beneficial for improving serum vitamin D levels, but their long-term use has unknown consequences.

The information obtained in this study will help in determining the efficacy of using a dietary supplement for improving serum vitamin D levels. By participating in the study, subjects may experience improved serum vitamin D level, bone formation, bone resorption, bone mineral density according to DEXA scan, flexibility, balance, and quality of life, while reducing their risk for other diseases. The risk of participating in this study is reasonable because the improvements in serum vitamin D level, bone formation, bone resorption, bone mineral density, flexibility, balance, gustatory response to the treatment, general inflammation, and quality of life associated with improved nutritional status will be enhanced.

The investigators are looking at an older population due to changes in all of our outcomes that are typically associated with aging. No consensus exists on what age is considered elderly, but the investigators have chosen 55 to have a wider age range. Other investigators have used non-elderly participants with a similar or higher dose of vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 55 years and over
* English or Spanish speaking
* Interest in participating in a novel nutritional supplement program
* Willingness to follow recommendations, including going off of all vitamin-D and calcium containing supplements, multivitamins, or OTC medications (e.g., Tums) 2 weeks before starting the study and during the intervention
* Scoring 0-2 errors on the Short Portable Mental Status Questionnaire

Exclusion Criteria:

* Less than 55 years of age
* Currently enrolled in another research trial for vitamin D dietary supplements or other bone disease treatments
* Unable to consent to the study
* Living in a skilled or intermediate care level nursing facility
* Women who are pregnant, during their period, or less than 2 days before or after their period at the time of the assessment
* Psychiatric diagnosis of schizophrenia, other psychotic disorders, bipolar disorder, major depression with psychotic features, delirium, and alcohol or substance abuse/dependence
* Bleeding disorders
* Aphasia or sensory, motor, and/or visual disturbances that could interfere with assessments, including inability to walk 10 feet without a walking aid
* Gastrointestinal disorders that could lead to uncertain resorption of the study supplements
* Major conditions such as neurologic, cardiovascular, pulmonary, renal, endocrine, thyroid, hepatic, autoimmune, or bone/joint that could interfere with vitamin D metabolism, psychometric tests, or body composition assessment (especially renal and heart failure)
* Erratic, accelerated, or mechanically-controlled irregular heart rhythms, atrial fibrillation/flutter, or atrioventricular block or implanted electronic device
* Any condition restricting blood flow, such as severe systemic vascular resistance
* Acute fever, diarrhea, or edema at the time of the assessment
* Dermatological lesions or excessive hair that would be in contact with the placement of the electrodes for the ESC assessment
* Hematologic or oncologic disorders treated with chemotherapy in the previous two years
* Dysfunctional levels of hemoglobins like carboxyhemoglobin or methemoglobin
* Active chemotherapy or radiation treatment for cancer
* Recent infusion of dyes into the bloodstream such as methylene blue, indocyanine green, indigo carmine, or fluorescein
* Diagnosis of a terminal illness
* Persons may not be in the second part of the study while participating in another trial for drugs, supplements, or treatment that affects serum vitamin D level
* Persons may not be in the second part of the study if they are unwilling to go off all vitamin D and calcium containing supplements, multivitamins, and over the counter medications 2 weeks prior to starting the study and for the duration of the second part of the study
* Persons may not be in this study if they are unwilling to have their blood drawn
* Persons may not be in the second part of the study if they are taking steroids, HCTZ, or any other drug known to interfere with vitamin D metabolism or taking diuretics or any other drug that interferes with hydration status
* Persons may not be in this study if they are unwilling to refrain from alcohol, caffeine, and stimulants (amphetamines) 12 hours before the examination
* Persons may not be in this study if they are unwilling to stop physical activity or sauna use 8 hours before the examination
* Persons may not be in this study if they are unwilling to remove fingernail polish or false fingernails during the testing

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Serum 25-(OH) D level at 6 months | Baseline, 6 months
  Vitamin D status defined by serum 25-(OH) D level. All serum measurements need to be taken in the morning following an overnight fast (before 9 AM).
Change from Baseline in Serum parathyroid hormone (PTH) levels at 6 months | Baseline, 6 months
  Serum parathyroid hormone (PTH) levels will be measured since serum 25 (OH) D levels corresponding to PTH inflection point are widely interpreted as a marker for vitamin D sufficiency. All serum measurements need to be taken in the morning following an overnight fast (before 9 AM).
Change from Baseline in Serum Osteocalcin at 6 months | Baseline, 6 months
  Bone formation as defined by serum osteocalcin. All serum measurements need to be taken in the morning following an overnight fast (before 9 AM).
Change from Baseline in Serum CTX at 6 months | Baseline, 6 months
  Bone resorption as defined by serum CTX. All serum measurements need to be taken in the morning following an overnight fast (before 9 AM).
Change from Baseline in Serum C-reactive Protein at 6 months | Baseline, 6 months
  General inflammation will be assessed by serum C-reactive protein; a key indicator of multiple inflammatory processes. All serum measurements need to be taken in the morning following an overnight fast (before 9 AM).

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 6 months | Baseline, 6 months
  Systolic blood pressure, diastolic blood pressure, and pulse will be measured to the nearest even digit by use of a random-zero sphygmomanometer (Mabis, IL, USA). Three readings will be made with the subjects seated after they have rested for five minutes. The average of the second and third readings will be used in the analysis.
Change from Baseline in Diastolic Blood Pressure at 6 months | Baseline, 6 months
  Systolic blood pressure, diastolic blood pressure, and pulse will be measured to the nearest even digit by use of a random-zero sphygmomanometer (Mabis, IL, USA). Three readings will be made with the subjects seated after they have rested for five minutes. The average of the second and third readings will be used in the analysis.
Pulse | Baseline, 6 months
  Systolic blood pressure, diastolic blood pressure, and pulse will be measured to the nearest even digit by use of a random-zero sphygmomanometer (Mabis, IL, USA). Three readings will be made with the subjects seated after they have rested for five minutes. The average of the second and third readings will be used in the analysis.
Change from Baseline in Gait Velocity at 6 months | Baseline, 6 months
  Dual task - Participants will be asked to perform the following tasks in a random order: usual walking (single task 1), counting backwards by 1 from 50 while standing (single task 2), and counting backwards by 1 from 50 while walking (dual task). Each participant's performance while walking during single and dual task test (without prioritizing either task) will be assessed by using the GAITRite portable electronic walkway system. The GAITRite system includes a 600 cm long and 64 cm wide walkway mat that is used to measure spatiotemporal gait parameters. The mat has imbedded sensors that are activated and deactivated according to foot pressure and is capable of measuring milliseconds and millimeters for time and length parameters, respectively. Before each trial participants will be given standardized instruction and a visual demonstration. The participants will be wearing comfortable, low-heeled shoes and will walk the length of the mat at the pace they select.
Change from Baseline in Step Length at 6 months | Baseline, 6 months
  Dual task - Participants will be asked to perform the following tasks in a random order: usual walking (single task 1), counting backwards by 1 from 50 while standing (single task 2), and counting backwards by 1 from 50 while walking (dual task). Each participant's performance while walking during single and dual task test (without prioritizing either task) will be assessed by using the GAITRite portable electronic walkway system. The GAITRite system includes a 600 cm long and 64 cm wide walkway mat that is used to measure spatiotemporal gait parameters. The mat has imbedded sensors that are activated and deactivated according to foot pressure and is capable of measuring milliseconds and millimeters for time and length parameters, respectively. Before each trial participants will be given standardized instruction and a visual demonstration. The participants will be wearing comfortable, low-heeled shoes and will walk the length of the mat at the pace they select.
Change from Baseline in Base of Support at 6 months | Baseline, 6 months
  Dual task - Participants will be asked to perform the following tasks in a random order: usual walking (single task 1), counting backwards by 1 from 50 while standing (single task 2), and counting backwards by 1 from 50 while walking (dual task). Each participant's performance while walking during single and dual task test (without prioritizing either task) will be assessed by using the GAITRite portable electronic walkway system. The GAITRite system includes a 600 cm long and 64 cm wide walkway mat that is used to measure spatiotemporal gait parameters. The mat has imbedded sensors that are activated and deactivated according to foot pressure and is capable of measuring milliseconds and millimeters for time and length parameters, respectively. Before each trial participants will be given standardized instruction and a visual demonstration. The participants will be wearing comfortable, low-heeled shoes and will walk the length of the mat at the pace they select.
Change from Baseline in Single Support Time at 6 months | Baseline, 6 months
  Dual task - Participants will be asked to perform the following tasks in a random order: usual walking (single task 1), counting backwards by 1 from 50 while standing (single task 2), and counting backwards by 1 from 50 while walking (dual task). Each participant's performance while walking during single and dual task test (without prioritizing either task) will be assessed by using the GAITRite portable electronic walkway system. The GAITRite system includes a 600 cm long and 64 cm wide walkway mat that is used to measure spatiotemporal gait parameters. The mat has imbedded sensors that are activated and deactivated according to foot pressure and is capable of measuring milliseconds and millimeters for time and length parameters, respectively. Before each trial participants will be given standardized instruction and a visual demonstration. The participants will be wearing comfortable, low-heeled shoes and will walk the length of the mat at the pace they select.
Change from Baseline in Double Support Time at 6 months | Baseline, 6 months
  Dual task - Participants will be asked to perform the following tasks in a random order: usual walking (single task 1), counting backwards by 1 from 50 while standing (single task 2), and counting backwards by 1 from 50 while walking (dual task). Each participant's performance while walking during single and dual task test (without prioritizing either task) will be assessed by using the GAITRite portable electronic walkway system. The GAITRite system includes a 600 cm long and 64 cm wide walkway mat that is used to measure spatiotemporal gait parameters. The mat has imbedded sensors that are activated and deactivated according to foot pressure and is capable of measuring milliseconds and millimeters for time and length parameters, respectively. Before each trial participants will be given standardized instruction and a visual demonstration. The participants will be wearing comfortable, low-heeled shoes and will walk the length of the mat at the pace they select.
Change from Baseline in Balance and Physical Performance at 6 months | Baseline, 6 months
  Balance and physical performance as measured with the Established Population for Epidemiologic Studies of the Elderly physical performance battery (EPESE), which includes: (a) side by side stands, (b) semi-tandem stand, (c) tandem stand, (d) measured walk, (e) repeated chair stands, and (f) timed chair stands.
Change from Baseline in Flexibility at 6 months | Baseline, 6 months
  Flexibility with the Sit and Reach Test will be assessed with the most common flexibility test by measuring the flexibility of the lower back and hamstrings. A box about 30 cm high and a meter rule is used to have the subject sit on the floor with his/her back straight. Legs are held straight ahead and knees flat against the floor. The box is placed flat against the feet (no shoes), and the arms are stretched out toward the box. The slide ruler on top of the box is positioned at the zero point. The subject leans forward slowly (without jerking or bouncing) as far as possible keeping the fingertips level with each other and the legs flat. The subject reaches slowly along the length of the ruler 3 times. On the third attempt, the subject reaches as far as possible and holds for 2 seconds and the score is recorded.
Change from Baseline in Physical Activity at 6 months | Baseline, 6 months
  Physical activity will be assessed with International Physical Activity Questionnaire (IPAQ). The IPAQ items are structured to provide individual domain specific scores for walking, moderate-intensity, and vigorous activity within the domains of work, transportation, domestic chores and gardening, and leisure-time. The tool asks about the time spent doing a specific physical activity in the last 7 days. For total scores, the duration (in minutes) and frequency for all types of activities in all domains are summed, while specific domain scores are calculated by the summation of the walking, moderate-intensity and vigorous-intensity activities within the specific domain. For activity-specific scores, the scores for the specific type of activity across domains are added. To measure the volume of activity, each type of activity is weighted by its energy requirement defined as the MET-min.
Change from Baseline in Vitamin D and Calcium intake at 6 months | Baseline, 6 months
  Vitamin D and Calcium intake will be assessed using a Vitamin D and Calcium Food Frequency Questionnaire. This tool allows estimation of the relative nutrient intakes based on foods eaten, frequency, and size. This short FFQ contains only 24 foods and beverages, and it is designed to assess vitamin D and calcium intake. The FFQ asks how frequently (never or less than once per month; 1/ month; 2-3/month; 1/week; 2/weeks; 3-4/week; 5-6/week; 1/day; 2-3/day) and how much of each of these foods is consumed based on medium serving size (small, medium, large). The short FFQ is associated with a database; therefore allowing the estimation of nutrient intakes for the reported portion size. Vitamin D and calcium values for the 24 foods will be recorded from the Diet History Questionnaire database developed by the National Cancer Institute, according to serving size.
Change from Baseline in Food Security at 6 months | Baseline, 6 months
  The 6-item U.S. Household Food Security Survey Module will be used to assess food security. The 6-item scale was developed by the National Center for Health Statistics. It asks the participant questions on foods eaten in the household in the last 12 months and whether they were able to afford the foods needed. Scores are coded as affirmative responses that are summed up to get a score. A score of 0-1 means high or marginal food security, 2-4 means low food security, and 5-6 means very low food security.
Change from Baseline in Sun Exposure at 6 months | Baseline, 6 months
  Sun Exposure Recall Questionnaire - Subjects' recollection of usual sun exposure over the previous year will be assessed via a questionnaire. This instrument measures the amount of time spent outdoors from 9 AM - 5 PM and amount of skin exposed for everyday of the week during summer and fall (June - December) and winter and spring (January - May), independently. This instrument also includes questions about sun protective behaviors including sunscreen and umbrella use. A scoring system is used to quantify time outdoors (<5 minutes; 5-30 minutes; and >30 min), sunscreen use, umbrella use, and amount of skin exposed (hands, face, arms, legs, bathing suit).
Change from Baseline in Quality of Life at 6 months | Baseline, 6 months
  The SF-36v2TM Health Survey provides psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure that does not target a specific age, disease, or treatment group.
Change from Baseline in Depression at 6 months | Baseline, 6 months
  Depression will be assessed using the Beck's depression questionnaire (BDI-II). It is a self-report 21 item instrument to assess the existence and severity of depressive symptoms. Each item corresponds to a symptom of depression and has a four-point scale ranging from 0 to 3, except for 2 items that have seven options to indicate decrease or increase in appetite and sleep. The score of all items are summed to give a single score. A total score of 0-13 is considered minimal, 14-19 mild, 20-28 moderate, and 29-63 severe.
Change from Baseline in Fear of Falling at 6 months | Baseline, 6 months
  Fall Efficacy Scale International (FES-I) is a 16-question assessment tool used to evaluate the fear of falling while performing activities like cleaning the house, getting dressed/undressed, preparing simple meals, taking a bath/shower, going to shop, getting in/out of the chair, going up/down stairs, walking around the neighborhood, reaching something above head/on ground, going to answer the phone before it stops ringing, walking on slippery surface, visiting friend/relative, walking in crowds, walking on uneven surfaces, walking up/down slope, and going out to a social event. The participants will be asked to rate on a scale of 1 to 4 how concerned they are about the possibility of falling while performing these activities with 1 meaning "not at all concerned," 2 being "somewhat concerned," 3 being "fairly concerned," and 4 being "very concerned."
Change from Baseline in Fall Frequency at 6 months | Baseline, 6 months
  History of falls will be assessed by asking the participant if they recall experiencing one or more falls in the last 6 months. A fall will be defined as an event that results in the person unintentionally coming to rest on the ground or other lower level with or without injury that is not due to a major intrinsic event, like seizure, stroke, loss of consciousness, epilepsy, excess alcohol, or an environmental hazard like sustaining a blow.
Change from Baseline in Compliance at 6 months | Baseline, 6 months
  Compliance will be measured using a modified version of the 8 item Morisky Medication Adherence Scale (MMAS-8). MMAS-8 is a generic self-report measure of medication taking behavior that does not target a specific age, disease, or treatment group.
Change from Baseline in Skin Color due to Sun Exposure at 6 months | Baseline, 6 months
  Reflectance colorimetry - Reflectance colorimetry using the IMS SmartProbe 400 will be used objectively measure sun exposure and skin color. This instrument measures the skin's reflectance of white light over a spectrum of wavelengths. The light is shined on the chosen area and the intensity of light reflected is measured by the probe. Melanin absorbs UV light; therefore, the more melanin present, and hence, the darker the skin, the less light is reflected back to the probe. The results are based on the Commission Internationale de l'Eclairage L scale endorsed by the International Commission on Illumination system as a way to represent accurately human color perception.

CONTACTS AND LOCATIONS:
Overall Officials: John Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Clinical Research Building, Miami, Florida, United States

REFERENCES:
- [Background] Chandra P, Binongo JN, Ziegler TR, Schlanger LE, Wang W, Someren JT, Tangpricha V. Cholecalciferol (vitamin D3) therapy and vitamin D insufficiency in patients with chronic kidney disease: a randomized controlled pilot study. Endocr Pract. 2008 Jan-Feb;14(1):10-7. doi: 10.4158/EP.14.1.10. PMID 18238736
- [Background] Vieth R, Chan PC, MacFarlane GD. Efficacy and safety of vitamin D3 intake exceeding the lowest observed adverse effect level. Am J Clin Nutr. 2001 Feb;73(2):288-94. doi: 10.1093/ajcn/73.2.288. PMID 11157326